CLINICAL TRIAL: NCT00202605
Title: A Phase II, Randomized, Double-Blind, Multi-center, Placebo-controlled, Crossover Study of SPD465 in Adults With Attention-Deficit Hyperactivity Disorder (ADHD)
Brief Title: Safety and Efficacy of SPD465 in Adults With ADHD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SPD465-203
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Amphetamine

INTERVENTIONS:
Drug: Neutral salts of dextroamphetamine sulfate, USP, amphetamine sulfate, USP, d-amphetamine saccharate, d,I-amphetamine aspartate monohydrate

SUMMARY:
The purpose of the study is to evaluate how safe and how well SPD465 works compared to placebo in adults with ADHD. It is hypothesized that SPD465 will achieve an extended duration of clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of ADHD using DSM-IV-TR criteria (at least 6 of the 9 subtype criteria met)
* Baseline ADHD-RS-IV score =>24
* IQ score of => 80 (using Kaufman Brief Intelligence Test)

Exclusion Criteria:

* BMI < 18.5 or > 30 kg/m2
* Diagnosis of Post Traumatic Stress Disorder, psychosis, bipolar illness, severe obsessive compulsive disorder, severe depressive or severe anxiety disorder
* History of seizure disorder or a lifetime history of any seizures (other than infantile febrile seizures), any tic disorder, or a current diagnosis and/or family history of Tourette's Disorder
* History of uncontrolled hypertension or currently hypertensive
* Subjects who have taken atomoxetine (STRATTERA) within 30 days prior to screening
* Current (or history within the last 12 months) of drug dependence or substance abuse disorder according to DSM-IV-TR criteria (excluding nicotine)
* Female subject is pregnant or lactating, less than 3 months post partum

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72
Dates: Start 2005-09-29 (Actual); Primary Completion 2006-01-06 (Actual); Study Completion 2006-01-06 (Actual)

PRIMARY OUTCOMES:
PERMP (Permanent Product Measure of Performance) | 0.5 hours pre-dosing
PERMP (Permanent Product Measure of Performance) | 2 hours post-dosing
PERMP (Permanent Product Measure of Performance) | 4 hours post-dosing
PERMP (Permanent Product Measure of Performance) | 8 hours post-dosing
PERMP (Permanent Product Measure of Performance) | 12 hours post-dosing
PERMP (Permanent Product Measure of Performance) | 14 hours post-dosing
PERMP (Permanent Product Measure of Performance) | 16 hours post-dosing

SECONDARY OUTCOMES:
Time Segment Rating System (ADHD-RS[TSRS]) | 5½, 11, and 16½ hours post-dosing
Subject self report (ADHD-SRS) of ADHD | approximately 5½, 11, and 16½ hours post-dosing
Treatment emergent adverse events | Throughout the study period of approximately 3.25 months.
Modified Pittsburgh Sleep Quality Index (PSQI) | Study orientation and randomization visit, Week 1 after Study orientation and randomization visit, Week 2 after Study orientation and randomization visit

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (4):
- United States (4):
  - Clinical Study Center, Little Rock, Arkansas
  - UCI Child Development Center, Irvine, California
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - Bayou City Research, Ltd., Houston, Texas

REFERENCES:
- [Derived] Wigal T, Childress A, Frick G, Yan B, Wigal S, Madhoo M. Effects of SHP465 mixed amphetamine salts in adults with ADHD in a simulated adult workplace environment. Postgrad Med. 2018 Jan;130(1):111-121. doi: 10.1080/00325481.2018.1389227. Epub 2017 Oct 31. PMID 29087231